CLINICAL TRIAL: NCT05377788
Title: Lazertinib Real-world Observational Study of in Pre-treated EGFR T790M Mutant With Advanced Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jin Seok Ahn, MD, Professor, Samsung Medical Center
Other Study IDs: KCSG LU22-01
Record Dates: First submitted 2022-05-04; First posted 2022-05-17 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; EGFR T790M
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — □Plasma Circulatory Tumor DNA Collection Blood: Before First Dose(laziertinib), End of Treatment(lazertinib) - Total 20ml (10ml*2 times)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective cohort: * Inclusion criteria
    * adults over the age of 19
    * Easter Cooperative Oncology Group performance 0-4
    * Patients who are eligible for or are being treated for test medication as per permit: patients with NSCLC with local progressive or metastatic EGFR T790M mutation who have previously been treated with Generation 1 or Generation 2 EGFR TKI
    * EGFR T790M mutation allows for all results identified in tumor tissue or plasma
    * Patients with brain MR within 3 months of study participation
  * After obtaining a consent form for research participation, follow-up and monitoring survival information and safety information. Survival follow-up of prospective cohorts will be followed up to the point of first occurrence during disease progression, withdrawal of consent, failure of follow-up investigation, and death.
  Interventions: Drug: Lazertinib
- Restrospective cohort: * Inclusion criteria
    * adults over the age of 19
    * Patients who are already using the lazertinib according to the domestic authorization of lazertinib(This includes when participants receive interventions as part of routine medical care)
  * Survival information is monitored after the time when the consent form for participation in the study is obtained. Survival follow-up of retrospective cohorts will be followed up to the point of first occurrence during disease progression, withdrawal of consent, failure of follow-up investigation, and death
  Interventions: Drug: Lazertinib

INTERVENTIONS:
Drug: Lazertinib — Treatment of EGFR T790M mutant-positive local progressive or metastatic non-small cell lung cancer patients who have previously been treated with EGFR
  Other Names: LECLAZA

SUMMARY:
* It is to evaluate the safety and effectiveness of a lasertinib(LECLAZA) single drug in a actual medical environment for patients

  1. Primary Purpose: Progression-free survival (PFS)
  2. Secondary Purpose:

     * Objective response rate
     * Time to treatment failure
     * Adverse event (AE), serious adverse event (SAE), and adverse event of special interest (AESI)
     * Severity of (S)AE
     * duration of response (DoR)
     * Overall survival (OS)
     * Intravenous Progressive Survival Period (Intracranial PFS)
     * Relative dose intensity
* Research Design : a Multi-Center Prospective and Restrospective Cohort Study

DETAILED DESCRIPTION:
□ the purpose of the study The study aims to explore the safety, efficacy and resistance of test drugs in patients with local progressive or metastatic epithelial growth factor T790M mutant non-small cell lung cancer who have been treated with epithelial growth factor receptor tyrosine kinase inhibitors.

This study is conducted in Korea. About 600 patients will be monitored until the first occurrence of disease progression, withdrawal of consent, failure of follow-up investigation, and death.

□ Research Procedures and Information Gathering Items There are no additional procedures performed by participating in this study and information on safety and effectiveness during the administration of Rexhraza will be followed up in routine care situations.

The information you will receive when you participate in this study is as follows.

* Subject characteristics, including age, gender, and race
* T790M Positive Mutation Status Results and Types of Tests Performed and Receptors
* a related medical history
* a physical examination
* disease characteristics
* history of chemotherapy
* associated concomitant medications
* administration of a test drug
* Safety and effectiveness
* Resistance mechanism in plasma circulation tumor DNA

ELIGIBILITY:
Inclusion Criteria:

1. Prospective cohort

   * adults over the age of 19
   * Easter Cooperative Oncology Group performance 0-4
   * Patients who are eligible for or are being treated for test medication as per permit: patients with NSCLC with local progressive or metastatic EGFR T790M mutation who have previously been treated with Generation 1 or Generation 2 EGFR TKI
   * EGFR T790M mutation allows for all results identified in tumor tissue or plasma
   * Patients with brain MR within 3 months of study participation
2. Rectrospective cohort

   * adults over the age of 19
   * Patients who are already using the test drug according to the domestic authorization of the test drug

Exclusion Criteria:

* Patients who have a history of hypersensitivity to test drugs or drugs of similar chemical structure or similar family to those of test drugs
* Pregnant women or lactating women
* Patients participating in other interventional clinical studies

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort: 300 people Prospective cohort: 600 people
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-07-31 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Through study completion, an average of 3 years
  Progression-free survival (PFS) is defined as the time from study enrollment until objective disease progression or death.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 3 years
  Objective response rate is defined as the proportion of patients who have a partial or complete response to therapy.
Time to treatment failure (TTF) | Through study completion, an average of 3 years
  Time to treatment failure (TTF) is defined as the interval between initiating therapy and the earliest of clinical progression, new locally directed or systemic treatment other than lazertinib.
Overall survival (OS) | Through study completion, an average of 3 years
  Overall survival (OS) is defined as the time from treatment to death.
Duration of response (DoR) | Through study completion, an average of 3 years
  Duration of response (DoR) is the length of time that a tumor continues to respond to treatment without cancer growing or spreading.
Intracranial Progression-free survival (Intracranial PFS) | Through study completion, an average of 3 years
  Intracranial PFS is defined as the time from study enrollment until objective intracranial progression.
Relative dose intensity | Through study completion, an average of 3 years
  Relative dose intensity is defined as the actual dose received divided by the standard calculated dose during a predefined period.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Seok Ahn, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn MJ, Han JY, Lee KH, Kim SW, Kim DW, Lee YG, Cho EK, Kim JH, Lee GW, Lee JS, Min YJ, Kim JS, Lee SS, Kim HR, Hong MH, Ahn JS, Sun JM, Kim HT, Lee DH, Kim S, Cho BC. Lazertinib in patients with EGFR mutation-positive advanced non-small-cell lung cancer: results from the dose escalation and dose expansion parts of a first-in-human, open-label, multicentre, phase 1-2 study. Lancet Oncol. 2019 Dec;20(12):1681-1690. doi: 10.1016/S1470-2045(19)30504-2. Epub 2019 Oct 3. PMID 31587882